CLINICAL TRIAL: NCT06375486
Title: A Single-arm, Single-center, Phase II Clinical Study of AK112 (a Dual-specific Antibody Against PD-1/VEGF) Combined With Hepatic Arterial Infusion Chemotherapy (HAIC) for the Treatment of Unresectable Hepatocellular Carcinoma.
Brief Title: Ivonescimab Combined With HAIC for the Treatment of Unresectable Hepatocellular Carcinoma（uHCC）.
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AK112-IIT-TianjinCIH-LHK
Record Dates: First submitted 2024-04-11; First posted 2024-04-19 (Actual); Last update posted 2024-04-19 (Actual); Status verified 2024-04

CONDITIONS: Hepatocellular Carcinoma Non-resectable; Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- AK112 arm (Experimental): The patients will receive AK112（PD-1/VEGF bispecific antibody）plus HAIC
  Interventions: Drug: Ivonescimab（AK112，a PD-1/VEGF bispecific antibody）

INTERVENTIONS:
Drug: Ivonescimab（AK112，a PD-1/VEGF bispecific antibody） — All enrolled subjects will receive Ivonescimab（AK112，a PD-1/VEGF bispecific antibody，20mg/kg Q3W) in combination with HAIC (utilizing the FOLFOX chemotherapy regimen)
  Other Names: HAIC

SUMMARY:
This study is a single-center, open-label Phase II clinical trial, aiming to enroll approximately 30 unresectable BCLC stage B or C hepatocellular carcinoma (HCC) patients from China. The primary objective is to evaluate the safety and efficacy of AK112 (a dual-specific antibody against PD-1/VEGF) in combination with hepatic arterial infusion chemotherapy (HAIC) for the treatment of unresectable hepatocellular carcinoma.

All enrolled subjects will receive AK112 (20mg/kg Q3W) combined with HAIC (utilizing the FOLFOX chemotherapy regimen) until the investigator determines no further clinical benefit (based on RECIST v1.1 imaging evaluation and clinical assessment), intolerable toxicity, completion of 24 months of treatment, or meeting other criteria for treatment discontinuation as outlined in the protocol, whichever occurs first.

DETAILED DESCRIPTION:
This study is a single-center, open-label Phase II clinical trial, planning to enroll approximately 30 Chinese subjects with unresectable BCLC stage B or C hepatocellular carcinoma (HCC). The primary objective is to evaluate the safety and efficacy of AK112 (a dual-specific antibody against PD-1/VEGF) in combination with hepatic arterial infusion chemotherapy (HAIC) for the treatment of unresectable hepatocellular carcinoma.

All enrolled subjects will receive AK112 (20mg/kg Q3W) in combination with HAIC (utilizing the FOLFOX chemotherapy regimen) until the investigator determines no further clinical benefit (based on RECIST v1.1 imaging assessment and clinical evaluation), intolerable toxicity, completion of 24 months of treatment, or meeting other criteria for treatment discontinuation as outlined in the protocol, whichever comes first.

The study consists of screening period (up to 28 days from subject signing informed consent form to the first dose), treatment period (including treatment visits during treatment and end-of-treatment visit), and follow-up period (including safety follow-up visits, disease progression follow-up visits, and survival follow-up). Subjects will undergo screening assessments within 28 days before the first dose to determine their eligibility for the study.

All subjects will undergo regular tumor response assessments, with objective response rate (ORR) evaluated by the investigator according to RECIST v1.1 and mRECIST criteria as the primary efficacy endpoint. Within the first 48 weeks after the initial dose, tumor assessments will be conducted every 6 weeks (±7 days), and after 48 weeks, assessments will be performed every 12 weeks (±7 days). If a subject discontinues study treatment for reasons other than disease progression or death, tumor assessments should continue according to a fixed schedule until radiographic progression or termination of study treatment (whichever occurs first), initiation of new anti-tumor therapy, loss to follow-up, death, withdrawal of informed consent, or study closure, whichever occurs first. Confirmation of objective response should occur at least 4 weeks after the initial documentation of response, and in cases of clinical stability, confirmation assessments can be performed at the next scheduled time point.

Adverse events (AEs) will be followed up to 30 days after the last dose or initiation of new anti-tumor therapy, whichever occurs first. Serious adverse events (SAEs) will be followed up to 90 days after the last dose or initiation of new anti-tumor therapy, whichever occurs first. Survival assessments will be conducted every 3 months after the last dose, and information on subsequent anti-tumor therapy will be collected after termination of study treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily sign a written informed consent form.
2. Age at enrollment is ≥ 18 years and ≤ 75 years, both males and females are eligible.
3. Eastern Cooperative Oncology Group (ECOG) performance status score of 0 or 1.
4. Expected survival ≥ 3 months.
5. Confirmed histologically/cytologically or cirrhotic patients meeting the Barcelona Clinic Liver Cancer (BCLC) stage B or C criteria for hepatocellular carcinoma (HCC) according to the American Association for the Study of Liver Diseases (AASLD) clinical diagnostic criteria.
6. Not suitable for curative treatment (surgery or ablation) and have not previously received systemic anti-tumor therapy for unresectable HCC.
7. Liver function classified as Child-Pugh class A.
8. Sufficient organ function.

Exclusion Criteria:

1. Components including fibrolamellar hepatocellular carcinoma, sarcomatoid hepatocellular carcinoma, cholangiocarcinoma, etc., confirmed histologically/cytologically.
2. Apart from HCC, subjects have had other malignant tumors within 5 years prior to enrollment. Subjects who have been cured of other malignant tumors through local treatment, such as basal or squamous cell carcinoma of the skin, superficial bladder cancer, cervical or breast carcinoma in situ, are not excluded. If diagnosed with liver cancer or other malignant tumors more than 5 years before dosing, pathological histology or cytology diagnosis of recurrent metastatic lesions is required.
3. Poor compliance, unable to cooperate and describe treatment responses.
4. History of past or current central nervous system (CNS) metastasis or leptomeningeal metastasis.
5. Presence of extrahepatic metastasis.
6. History of hepatic encephalopathy or liver transplantation.
7. Clinical symptoms or recurrent pleural effusion, pericardial effusion, or ascites requiring repeated drainage.
8. Currently participating in interventional clinical research treatment, or have received other investigational drugs or used investigational devices within 4 weeks prior to the first dose.
9. History of or current non-infectious pneumonia or interstitial lung disease requiring systemic corticosteroid therapy.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-03-14 (Actual); Primary Completion 2025-03-14 (Estimated); Study Completion 2026-06-15 (Estimated)

PRIMARY OUTCOMES:
Overall response rate (ORR) | up to 1 year
  Defined as proportion of patients who have a best response of CR or PR

SECONDARY OUTCOMES:
Progress Free Survival （PFS） | up to 2 years
  Defined as the time from enrollment to disease progression or death (whichever occurs first)
Overall survival (OS) | up to 2 years
  OS is defined as the time from date of neoadjuvant treatment start to the date of death from any cause or to the date of last follow-up if patients are alive. If a patient is alive by the time of final analysis, the patient will be censored at the last follow-up date.
Adverse Events（AEs） | up to 3 years
  Defined as the proportion of patients with AE, treatment-related AE (TRAE), immune-related AE (irAE), serious adverse event (SAE), assessed by NCI CTCAE v5.0

CONTACTS AND LOCATIONS:
Locations (1):
- Tianjin Cancer Hospital Airport Hospital, Tianjin, Tianjin Municipality, China